CLINICAL TRIAL: NCT05873504
Title: Outcome Comparisons of Two Vibratory Positive Expiratory Pressure Devices in Patients Unable to Clear Airway Secretions
Brief Title: Outcome Comparisons of Vibratory Airway Clearance Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23011705
Record Dates: First submitted 2023-04-16; First posted 2023-05-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Airway Clearance Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Oscillatory Index Device (Experimental): Patients in this arm will receive a device that vibrates with high oscillatory index.
  Interventions: Device: High Oscillatory Index Device
- Low Oscillatory Index Device (Active Comparator): Patients in this arm will receive a device that vibrates with low oscillatory index.
  Interventions: Device: Low Oscillatory Index Device

INTERVENTIONS:
Device: High Oscillatory Index Device — This device is commonly used to provide assistance with airway secretion clearance.
  Other Names: Aerobika
  Arms: High Oscillatory Index Device
Device: Low Oscillatory Index Device — This device is commonly used to provide assistance with airway secretion clearance.
  Other Names: VibraPEP
  Arms: Low Oscillatory Index Device

SUMMARY:
This pilot study aims to compare the ability of a higher oscillatory index device versus a lower oscillatory index device on airway secretion clearance and other clinically significant outcomes.

DETAILED DESCRIPTION:
This pilot study is a randomized control trial of adult patients admitted to an academic medical center. Subjects included in this study must be adults 18 years or older and will receive a respiratory assessment and allocation of therapy (RAAT) score of at least 10 and a secretion score of at least 5. Exclusion criteria include those younger than 18 years of age, those who are pregnant, with an SVC of <10mL/kg, and who cannot follow instructions or currently receiving cough assist, vest or intrapulmonary percussive ventilation. Patients receiving more than one therapy session using the oscillatory index device before enrollment will be excluded. Patients with multiple ICU admissions will be enrolled once. After randomization, the study team will give the device to the patient and administer instructions on the device use. Each eligible patient will receive clinical evaluation using RAAT scores per the department policy. The frequency of using oscillatory index devices will be based on the department protocol. Each subject will be followed up until discharge from the hospital. The primary outcome will be the RAAT score. The RAAT score range from 0-50 and includes five components: respiratory rate, oxygen therapy, chest x-ray, secretion clearance, and vital capacity. The higher score denotes respiratory compromise, and therapy is assigned for score 10 or greater per departmental protocol. The secondary outcomes include respiratory interventions used or other bronchial hygiene (vest therapy, intrapulmonary percussive ventilation) performed, ICU re-admission, need for continuous positive pressure, and length of stay (hospital and ICU).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Respiratory assess and treat (RAAT) score of at least 10 and a secretion score of at least 5

Exclusion Criteria:

* Younger than 18 years of age
* Pregnant
* Slow vital capacity (SVC) of <10 mL/kg
* Unable to follow instructions
* Currently receiving cough assist, vest therapy or intrapulmonary percussive ventilation
* Received more than 1 therapy session using oscillatory index device
* Multiple ICU admission with previous study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory assess and treat (RAAT) score | Change from baseline RAAT score at 12 hours
  The RAAT score range from 0-50.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT05873504/ICF_001.pdf